CLINICAL TRIAL: NCT03314805
Title: PG2 Treatment for Reduction of Chemotherapy-Induced Toxicity and Encouraging Compliance With Chemotherapy Among Stage II/III Breast Cancer Patients Receiving Adjuvant Chemotherapy
Brief Title: PG2 Treatment Among Stage II/III Breast Cancer Patients Receiving Adjuvant Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PH-CP026
Record Dates: First submitted 2017-09-26; First posted 2017-10-19 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Cancer-related Fatigue; Neutropenia, Malignant
Keywords: astragalus polysaccharides; breast cancer; adjuvant chemotherapy
MeSH Terms: conditions — Acquired agranulocytosis; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Procedure: EC Chemotherapy
- Treatment (Experimental): Astragalus polysaccharides 500 mg
  Interventions: Drug: Astragalus polysaccharides 500 mg; Procedure: EC Chemotherapy

INTERVENTIONS:
Drug: Astragalus polysaccharides 500 mg — PG2 (500 mg in 500 ml saline), 3 days via i.v. infusion per chemotherapy cycle
  Other Names: PG2 Lyo. Injection 500 mg
  Arms: Treatment
Drug: Placebo — 500 ml saline, 3 days via i.v. infusion per chemotherapy cycle
  Arms: Control
Procedure: EC Chemotherapy — Epirubicin plus Cyclophosphamide every 21 days

SUMMARY:
Adjuvant chemotherapy usually is recommended after surgery for breast cancer patients who are at significant risk for disseminated disease. Chemotherapy has been demonstrated to reduce the risk of breast cancer recurrence. Anthracycline-based regimens, including doxorubin or epilubicin, are the breast cancer adjuvant chemotherapy standards of care. Fatigue has also been identified as the most problem for breast cancer patients under adjuvant chemotherapy. In the current study, it is aimed to show that PG2 (astragalus polysaccharides) treatment among stage II/III breast patients under adjuvant EC regimen in reduction of chemotherapy-induced toxicity and encouraging compliance with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Women who are able to provide informed consent
* Age 20 years and older
* Diagnosis of stage II to III breast cancer
* Patients who had undergone surgery for breast cancer treatment.
* Planning to receive anthracycline -based adjuvant chemotherapy
* Have adequate bone marrow, liver, and renal function
* ECOG ≦1
* Willing and able to complete quality of life questionnaires.

Exclusion Criteria:

* Pregnancy or lactating women.
* Baseline BFI score >3.
* History of chronic fatigue syndrome, uncontrolled active infection, active cardiac disease, poor controlled hypertension or diabetes mellitus, any serious medical condition, psychiatric illness, and regular steroid therapy as determined by investigators.
* History of previous breast cancer or other malignancy within the past 3 years with the exception of adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer.
* Known severe allergy to Astragalus membranaceus or its mayor extracts (polysaccharides).

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 67 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Change in chemotherapy-related fatigue by brief fatigue Inventory | through 4 chemotherapy cycles (each cycle is 21 days)
Incidence of Grade 3/4 neutropenia | through 4 chemotherapy cycles (each cycle is 21 days)

SECONDARY OUTCOMES:
Incidence of other Grade 3/4 Hematologic Toxicities | through study completion, an average 6-8 chemotherapy cycles (each cycle is 21 days)
Chemotherapy Dose Reductions | through study completion, an average 6-8 chemotherapy cycles (each cycle is 21 days)
Days of chemotherapy delay | through study completion, an average 6-8 chemotherapy cycles (each cycle is 21 days)
Cumulative Doses of G-CSF consumption | through study completion, an average 6-8 chemotherapy cycles (each cycle is 21 days)
Health-related Quality of Life by EORTC QLQ-C30 & Br23 | through study completion, an average 6-8 chemotherapy cycles (each cycle is 21 days)
ECOG | through study completion, an average 6-8 chemotherapy cycles (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ming Rau, MD, Principal Investigator — E-Da Cancer Hospital
Locations (5):
- Taiwan (5):
  - E-Da Cancer Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Kaohsiung Branch, Kaohsiung City
  - Chang Gung Memorial Hospital, Lovers Lake branch, Keelung
  - Chang Gung Memorial Hospital, Taipei Branch, Taipei
  - Chang Gung Memorial Hospital, Linkou Branch, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen WC, Chen SC, Wang CH, Hung CM, Peng MT, Liu CT, Chang YS, Kuo WL, Chou HH, Yeh KY, Wu TH, Wu CF, Chang PH, Huang YM, Yu CC, Lee CH, Rau KM. Astragalus polysaccharides improve adjuvant chemotherapy-induced fatigue for patients with early breast cancer. Sci Rep. 2024 Oct 28;14(1):25690. doi: 10.1038/s41598-024-76627-z. PMID 39465324